CLINICAL TRIAL: NCT03760653
Title: Physical Activity Along With a Probiotic for the Immune System and Quality of Life Improvement in Breast Cancer Survivor: A Randomised Controlled Pilot Study
Brief Title: Synergic Effects of Physical Activity and Probiotic on Gut Immune System and Quality of Life of Breast Cancer Survivors.
Acronym: ESICA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The researcher who was able to recruit the patients abandoned the project.
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Mar Larrosa, Senior Researcher, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UEM0002
Record Dates: First submitted 2018-11-07; First posted 2018-11-30 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer Females
Keywords: Breast Cancer Survivor; Probiotic; Immune System; Physical Exercise; Quality of Life; Gut Microbiota
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The probiotic and the placebo will be encapsulated in identical capsules and in identical cans that will only be identified with the letters A and B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Physical Exercise and probiotic group (Experimental): The subjects will receive 3 weekly sessions of combined exercise supervised by professionals in a specialized gym (60 minutes each one). The exercise will consist of a combination of aerobic and strength exercises involving the main muscle groups. They will take the probiotic supplementation at the established dose, 3 capsules/day before bedtime. Each probiotic capsule contains Lactobacillus rhamnosus, Lactobacillus paracasei, Lactobacillus acidophilus, Bifidobacterium bifidum.
  Interventions: Other: Physical Exercise and probiotic group
- Probiotic group (Experimental): Participants will follow their usual sedentary lifestyle (i.e to practice less than 3 days a week of physical exercise, as is specified in the inclusion criteria). They will take the probiotic supplementation at the established dose. Each probiotic capsule contains Lactobacillus rhamnosus, Lactobacillus paracasei, Lactobacillus acidophilus, Bifidobacterium bifidum
  Interventions: Dietary Supplement: Probiotic group
- Placebo group (Placebo Comparator): They will follow their sedentary lifestyle. Placebo probiotic will consist of a maltodextrin capsule.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Other: Physical Exercise and probiotic group — The exercise intervention will last 12 weeks. It will include three weekly sessions of programmed physical exercise of ~ 60 min duration (aerobic and strength combined training). The exercise sessions will be individualized and will follow the rules of the world reference institutions for aerobic training. Each session will be held in a authorized fitness center and it will be supervised and individualized for each subject by expert professionals.The probiotic will be taken (3 capsules/day) for 12 weeks. Each probiotic capsule contains Lactobacillus rhamnosus, Lactobacillus paracasei, Lactobacillus acidophilus, Bifidobacterium bifidum.
  Arms: Physical Exercise and probiotic group
Dietary Supplement: Probiotic group — Probiotic supplementation (3 capsules/day) will be taken before bedtime for 12 weeks.Each probiotic capsule contains Lactobacillus rhamnosus, Lactobacillus paracasei, Lactobacillus acidophilus, Bifidobacterium bifidum.
  Arms: Probiotic group
Dietary Supplement: Placebo group — Subjects will take 3 capsules/day of placebo capsules (maltodextrin) for 12 weeks
  Arms: Placebo group

SUMMARY:
Physical exercise along with gut microbiota improvement -because of probiotic intake- can improve the quality of life and immune system in breast cancer survivors. This is achieved because exercise improves the muscle mass in cancer patients (often reduced by treatment and/or inactivity), together with the gut microbiota improvement, this stimulates the inmune system function, improving the quality of life of these patients.

DETAILED DESCRIPTION:
The aim of this study is to determine the effects of physical exercise together with the supplementation of a probiotic on gut microbiota balance, the gut immune system and quality of life (intended as functional and muscular capacity, physical qualities and emotional state) in breast cancer survivors .

A randomized controlled pilot study has been designed in three parallel groups. Breast cancer survivors will be randomly assigned to each of the 3 groups: a) probiotic supplementation + supervised combined physical exercise (PEF), b) probiotic supplementation and habitual sedentary lifestyle (P), and c) control group will follow their usual lifestyle and will receive a placebo (C).

The exercise intervention will last 12 weeks. It will include three weekly sessions of programmed physical exercise of ~ 60 min duration (combined training). The exercise program will be individualized and will follow the rules of the world reference institutions for aerobic training. Each session will be held in a qualified fitness center and it will be supervised and individualized for each subject by professional experts .The two supplemented groups will take 3 capsules (Lactobacillus rhamnosus, Lactobacillus paracasei, Lactobacillus acidophilus, Bifidobacterium bifidum) a day (at night before bedtime) for 12 weeks.

The variables gut microbiota, fecal levels of immunoglobulin A, cardiorespiratory capacity, anthropometry variables, lifestyle, muscular capacity, quality of life, anxiety, depression and stress levels will be analized at the beginning (baseline dose) and after 12 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Breast Cancer Survivors
* <18 aged.
* No chemotherapy treatment or that at least three months have passed after the last chemotherapy treatment before the beginning of the study.
* Breast cancer status: I-IV status.
* ECOG scale: 0-1.
* Normal weight.

Exclusion Criteria:

* Extreme Diet.
* Exercise practice (at least at the doses recommended by WHO)
* Presence of heart disease
* Uncontrolled blood hypertension: (>160/90 mmHg).
* Uncontrolled metabolic disease
* Infectious chronic disease
* Uncontrolled pain
* Pregnancy or breast feeding
* Gastrointestinal disease
* Alcoholism
* Any condition that contraindicates the exercise practice in survivors cancer (fractures risk, severe leukopenia , low platelet count)
* Antibiotics intake during the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer survivors
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life of breast cancer survivors | Quality of life will be analyzed at the beginning (baseline dose) and after 12 weeks of intervention
  Breast cancer survivors quality of life will be analyzed with the quality of life questionnaire from The European Organization for Research and Treatment of Cancer EORTC QLQ BR-23 test (a specific module for breast cancer survivors)

SECONDARY OUTCOMES:
Change in Functional capacity | Functional capacity and physical quality will be analyzed at the beginning (baseline dose) and after 12 weeks of exercise intervention
  Dynamic fitness cardiorespiratory
Change in Body Composition | Functional capacity and physical quality will be analyzed at the beginning (baseline dose) and after 12 weeks of exercise intervention
  Body Mass Index
Change in Muscular Capacity | Muscular capacity will be analyzed at the beginning (baseline dose) and after 12 weeks of intervention.
  Pressure manual test will be determined
Change in Dietary habits | Lifestyle will be analyzed at the beginning (baseline dose) and after 12 weeks of intervention
  Food Frequency Questionnaire
Change in Physical activity level | Lifestyle will be analyzed at the beginning (baseline dose) and after 12 weeks of intervention
  Physical activity questionnaire (IPAQ) will be used
Change in Anxiety state | Emotional state will be analyzed at the beginning (baseline dose) and after 12 weeks of intervention
  The State-Trait Anxiety Inventory (STAI)
Change in Depression state | Emotional state will be analyzed at the beginning (baseline dose) and after 12 weeks of intervention
  Depression inventory (IDER)
Change Stress state | Emotional state will be analyzed at the beginning (baseline dose) and after 12 weeks of intervention
  Stress coping questionnarie for oncology patients will be used
Change in Gut Microbiota | Gut microbiota will be analyzed at the beginning (baseline dose) and after 12 weeks of intervention)
  Microbial diversity, bifidobacteria and lactobacillus percentage
Change in Immune system | Immunoglobulin A levels will be analyzed at the beginning (baseline dose) and after 12 weeks of intervention
  Fecal immunoglobulin A levels

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Herrero, PhD, Study Director — Centro medicina deportiva Miranda Ebro
Locations (1):
- Mar Larrosa, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Battaglini CL, Mills RC, Phillips BL, Lee JT, Story CE, Nascimento MG, Hackney AC. Twenty-five years of research on the effects of exercise training in breast cancer survivors: A systematic review of the literature. World J Clin Oncol. 2014 May 10;5(2):177-90. doi: 10.5306/wjco.v5.i2.177. PMID 24829866
- [Background] Benton MJ, Schlairet MC, Gibson DR. Change in quality of life among breast cancer survivors after resistance training: is there an effect of age? J Aging Phys Act. 2014 Apr;22(2):178-85. doi: 10.1123/japa.2012-0227. Epub 2013 Apr 9. PMID 23579251
- [Background] Bressa C, Bailen-Andrino M, Perez-Santiago J, Gonzalez-Soltero R, Perez M, Montalvo-Lominchar MG, Mate-Munoz JL, Dominguez R, Moreno D, Larrosa M. Differences in gut microbiota profile between women with active lifestyle and sedentary women. PLoS One. 2017 Feb 10;12(2):e0171352. doi: 10.1371/journal.pone.0171352. eCollection 2017. PMID 28187199
- [Background] Campbell KL, Pusic AL, Zucker DS, McNeely ML, Binkley JM, Cheville AL, Harwood KJ. A prospective model of care for breast cancer rehabilitation: function. Cancer. 2012 Apr 15;118(8 Suppl):2300-11. doi: 10.1002/cncr.27464. PMID 22488704
- [Background] Cerda B, Perez M, Perez-Santiago JD, Tornero-Aguilera JF, Gonzalez-Soltero R, Larrosa M. Gut Microbiota Modification: Another Piece in the Puzzle of the Benefits of Physical Exercise in Health? Front Physiol. 2016 Feb 18;7:51. doi: 10.3389/fphys.2016.00051. eCollection 2016. PMID 26924990
- [Background] Cramp F, Byron-Daniel J. Exercise for the management of cancer-related fatigue in adults. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD006145. doi: 10.1002/14651858.CD006145.pub3. PMID 23152233
- [Background] Dulko D, Pace CM, Dittus KL, Sprague BL, Pollack LA, Hawkins NA, Geller BM. Barriers and facilitators to implementing cancer survivorship care plans. Oncol Nurs Forum. 2013 Nov;40(6):575-80. doi: 10.1188/13.ONF.575-580. PMID 24161636
- [Background] Erdman SE, Poutahidis T. Gut bacteria and cancer. Biochim Biophys Acta. 2015 Aug;1856(1):86-90. doi: 10.1016/j.bbcan.2015.05.007. Epub 2015 Jun 4. PMID 26050963
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Fong DY, Ho JW, Hui BP, Lee AM, Macfarlane DJ, Leung SS, Cerin E, Chan WY, Leung IP, Lam SH, Taylor AJ, Cheng KK. Physical activity for cancer survivors: meta-analysis of randomised controlled trials. BMJ. 2012 Jan 30;344:e70. doi: 10.1136/bmj.e70. PMID 22294757
- [Background] Forsythe LP, Alfano CM, George SM, McTiernan A, Baumgartner KB, Bernstein L, Ballard-Barbash R. Pain in long-term breast cancer survivors: the role of body mass index, physical activity, and sedentary behavior. Breast Cancer Res Treat. 2013 Jan;137(2):617-30. doi: 10.1007/s10549-012-2335-7. Epub 2012 Dec 15. PMID 23242613
- [Background] Gnagnarella P, Draga D, Baggi F, Simoncini MC, Sabbatini A, Mazzocco K, Bassi FD, Pravettoni G, Maisonneuve P. Promoting weight loss through diet and exercise in overweight or obese breast cancer survivors (InForma): study protocol for a randomized controlled trial. Trials. 2016 Jul 28;17:363. doi: 10.1186/s13063-016-1487-x. PMID 27464488
- [Background] Hallal PC, Victora CG. Reliability and validity of the International Physical Activity Questionnaire (IPAQ). Med Sci Sports Exerc. 2004 Mar;36(3):556. doi: 10.1249/01.mss.0000117161.66394.07. No abstract available. PMID 15076800
- [Background] Goedert JJ, Jones G, Hua X, Xu X, Yu G, Flores R, Falk RT, Gail MH, Shi J, Ravel J, Feigelson HS. Investigation of the association between the fecal microbiota and breast cancer in postmenopausal women: a population-based case-control pilot study. J Natl Cancer Inst. 2015 Jun 1;107(8):djv147. doi: 10.1093/jnci/djv147. Print 2015 Aug. PMID 26032724
- [Background] Herrero F, San Juan AF, Fleck SJ, Balmer J, Perez M, Canete S, Earnest CP, Foster C, Lucia A. Combined aerobic and resistance training in breast cancer survivors: A randomized, controlled pilot trial. Int J Sports Med. 2006 Jul;27(7):573-80. doi: 10.1055/s-2005-865848. PMID 16802254
- [Background] Lozupone C, Knight R. UniFrac: a new phylogenetic method for comparing microbial communities. Appl Environ Microbiol. 2005 Dec;71(12):8228-35. doi: 10.1128/AEM.71.12.8228-8235.2005. PMID 16332807
- [Background] Minton O, Berger A, Barsevick A, Cramp F, Goedendorp M, Mitchell SA, Stone PC. Cancer-related fatigue and its impact on functioning. Cancer. 2013 Jun 1;119 Suppl 11:2124-30. doi: 10.1002/cncr.28058. PMID 23695924
- [Background] Mirandola D, Miccinesi G, Muraca MG, Sgambati E, Monaci M, Marini M. Evidence for adapted physical activity as an effective intervention for upper limb mobility and quality of life in breast cancer survivors. J Phys Act Health. 2014 May;11(4):814-22. doi: 10.1123/jpah.2012-0119. Epub 2013 Apr 5. PMID 23575310
- [Background] Mukaida N. Intestinal microbiota: unexpected alliance with tumor therapy. Immunotherapy. 2014;6(3):231-3. doi: 10.2217/imt.13.170. PMID 24762069
- [Background] Phillips SM, Dodd KW, Steeves J, McClain J, Alfano CM, McAuley E. Physical activity and sedentary behavior in breast cancer survivors: New insight into activity patterns and potential intervention targets. Gynecol Oncol. 2015 Aug;138(2):398-404. doi: 10.1016/j.ygyno.2015.05.026. Epub 2015 May 28. PMID 26026737
- [Background] Rao VP, Poutahidis T, Ge Z, Nambiar PR, Boussahmain C, Wang YY, Horwitz BH, Fox JG, Erdman SE. Innate immune inflammatory response against enteric bacteria Helicobacter hepaticus induces mammary adenocarcinoma in mice. Cancer Res. 2006 Aug 1;66(15):7395-400. doi: 10.1158/0008-5472.CAN-06-0558. PMID 16885333
- [Background] Rogers LQ, Courneya KS, Anton PM, Verhulst S, Vicari SK, Robbs RS, McAuley E. Effects of a multicomponent physical activity behavior change intervention on fatigue, anxiety, and depressive symptomatology in breast cancer survivors: randomized trial. Psychooncology. 2017 Nov;26(11):1901-1906. doi: 10.1002/pon.4254. Epub 2016 Sep 6. PMID 27530961
- [Background] Saad R, Rizkallah MR, Aziz RK. Gut Pharmacomicrobiomics: the tip of an iceberg of complex interactions between drugs and gut-associated microbes. Gut Pathog. 2012 Nov 30;4(1):16. doi: 10.1186/1757-4749-4-16. PMID 23194438
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Travier N, Fonseca-Nunes A, Javierre C, Guillamo E, Arribas L, Peiro I, Buckland G, Moreno F, Urruticoechea A, Oviedo GR, Roca A, Hurtos L, Ortega V, Munoz M, Garrigos L, Cirauqui B, Del Barco S, Arcusa A, Segui MA, Borras JM, Gonzalez CA, Agudo A. Effect of a diet and physical activity intervention on body weight and nutritional patterns in overweight and obese breast cancer survivors. Med Oncol. 2014 Jan;31(1):783. doi: 10.1007/s12032-013-0783-5. Epub 2013 Dec 6. PMID 24310809
- [Background] Travier N, Guillamo E, Oviedo GR, Valls J, Buckland G, Fonseca-Nunes A, Alamo JM, Arribas L, Moreno F, Sanz TE, Borras JM, Agudo A, Javierre C. Is Quality of Life Related to Cardiorespiratory Fitness in Overweight and Obese Breast Cancer Survivors? Women Health. 2015;55(5):505-24. doi: 10.1080/03630242.2015.1022817. Epub 2015 Apr 2. PMID 25833659
- [Background] van Vliet MJ, Harmsen HJ, de Bont ES, Tissing WJ. The role of intestinal microbiota in the development and severity of chemotherapy-induced mucositis. PLoS Pathog. 2010 May 27;6(5):e1000879. doi: 10.1371/journal.ppat.1000879. PMID 20523891
- [Background] Viaud S, Daillere R, Boneca IG, Lepage P, Langella P, Chamaillard M, Pittet MJ, Ghiringhelli F, Trinchieri G, Goldszmid R, Zitvogel L. Gut microbiome and anticancer immune response: really hot Sh*t! Cell Death Differ. 2015 Feb;22(2):199-214. doi: 10.1038/cdd.2014.56. Epub 2014 May 16. PMID 24832470